CLINICAL TRIAL: NCT00652561
Title: An Open-Label, Non-Randomized, Multicenter, Three Stage, Phase 2 Study of S-1 as 2nd Line Therapy for Patients With Advanced Non-Small Cell Lung Cancer (Stage IIIB/Stage IV)
Brief Title: Phase 2 Study of S-1 as 2nd Line Therapy in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry); United BioSource, LLC (Industry)
Responsible Party: Fabio Benedetti, M.D., Chief Medical Officer, Taiho Pharma USA, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1203; NCT00227552 (obsolete NCT alias)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All patients will receive S-1 orally at a dose of 30 mg/m2 twice daily (BID) for 14 days followed by a 1-week recovery period, repeated every 3 weeks.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — All patients will receive S-1 orally at a dose of 30 mg/m2 twice daily (BID) for 14 days followed by a 1-week recovery period, repeated every 3 weeks. The study may go to the second stage only if the stage 2 criteria are met, where 3/30 (10%) or more patients must have achieved a confirmed response (CR or PR) in stage 1.The study may go to the third stage only if at least 8/50 patients (16%) must have achieved a confirmed response in stage 2

SUMMARY:
The purpose of this study is to determine whether S-1 is effective as 2nd line therapy in slowing tumor activity in patients with advanced non-small cell lung cancer. The study is also looking at the safety of S-1.

DETAILED DESCRIPTION:
Advanced non-small cell lung cancer is relatively unresponsive to chemotherapy. This is true for the nucleoside analogue gemcitabine, with a response rate of approximately 10%, as well as for 5-fluorouracil (5-FU). Even when gemcitabine is combined with other chemotherapeutic drugs or biological agents, the overall tumor response rate remains basically unchanged. S-1 is a new generation oral fluoropyrimidine that combines Tegafur (5-fluoro-1-(tetrahydro-2-furanyl)-2,4(1H,3H)-pyrimidinedione [FT]), an oral prodrug of 5-FU, with two modulators, Gimeracil (5-chloro-2,4-dihydroxypyridine [CDHP]), which inhibits 5-FU degradation by dihydropyrimidine dehydrogenase (DPD) inhibition, and Oteracil potassium (Oxo), which inhibits 5-FU phosphorylation in the digestive tract. This combination of 3 compounds is designed to achieve enhanced antitumor activity while decreasing gastrointestinal toxicity.

This is an open-label, multicenter, single-arm, 3-stage, Phase 2 study evaluating the efficacy and safety of single agent S-1 as 2nd line therapy for patients with advanced NSCLC. The 3 stages of this study correspond to a futility stage (stage 1), a decision stage (stage 2), and a stage for improvement of precision of ORR (stage 3).

ELIGIBILITY:
Inclusion Criteria:

* 1. Has given written informed consent. 2. Has histologically and/or cytologically proven unresectable or recurrent NSCLC stage IIIB with pleural effusion or pericardial effusion, or stage IV (mixed forms with small cell lung cancer are excluded).

  3. Has received prior 1st line chemotherapy combination (platinum or non-platinum-based) treatment and has not received any 2nd line therapy.

  4. Has measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, ie, has at least one measurable lesion. A measurable lesion is one that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm using spiral Computed Tomography (CT) scan.

  5. Is able to take medications orally. 6. Is ≥ 18 years of age. 7. Has an ECOG performance status 0 or 1. 8. Has adequate organ function as defined by the following criteria:
  1. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN; if liver function abnormalities are due to underlying liver metastasis AST (SGOT) and ALT (SGPT) ≤ 5 x ULN.
  2. Total serum bilirubin of ≤ 1.5 x ULN.
  3. Absolute granulocyte count of ≥ 1,500/mm3.
  4. Platelet count ≥ 100,000/mm3.
  5. Hemoglobin of ≥ 9.0 g/dL.
  6. Calculated creatinine clearance (CrCl) ≥ 60 mL/min (Cockcroft-Gault formula). 9. Is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

     Exclusion Criteria:
* 1. Has had treatment with any of the following within the specified time frame prior to study drug administration:

  1. Any investigational agent either concurrently or within the past 30 days.
  2. Any prior 1st line treatment with S-1 for NSCLC.
  3. Previous therapy for NSCLC within the past 21 days, including any chemotherapy, immunotherapy, biologic or hormonal therapy (6 weeks for nitrosureas or mitomycin C).
  4. Radiotherapy within the prior 2 weeks.
  5. Any radiation therapy to a target lesion within the past 3 months, unless there was evidence of PD after radiotherapy (and this target lesion must not be the only site of measurable disease).
  6. Current enrollment in another clinical study with an investigational agent. Patients participating in surveys or observational studies are eligible to participate in this study.

     2. Has a serious illness or medical condition(s) including, but not limited to, the following:

  <!-- -->

  1. Other active malignancies.
  2. Symptomatic brain metastasis not controlled by corticosteroids.
  3. Leptomeningeal metastasis.
  4. Myocardial infarction within the last 6 months, severe/unstable angina, congestive heart failure New York Heart Association (NYHA) class III or IV.
  5. Chronic nausea, vomiting, and/or diarrhea.
  6. Psychiatric disorder that may interfere with consent and/or protocol compliance.
  7. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
  8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.

     3. Is receiving concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1:

  <!-- -->

  1. Sorivudine, uracil, cimetidine, folinic acid, and dipyridamole (may enhance S-1 activity).
  2. Allopurinol (may diminish S-1 activity).
  3. Phenytoin (S-1 may enhance phenytoin activity).
  4. Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 activity).

     4. Is a pregnant or lactating female. 5. With reproductive potential and refuses to use an adequate means of contraception (including male patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Overall tumor response rate (ORR - the proportion of patients with objective evidence of PR or CR) | Each cycle will last 21 days (14 days treatment, 7 days recovery) until death or removal from study for any reason. Tumor assessmentswill be obtained at baseline and at the end of every even cycle

SECONDARY OUTCOMES:
To evaluate the duration of response (DR), and progression-free survival (PFS) | Each cycle will last 21 days (14 days treatment, 7 days recovery) until death or removal from study for any reason. Pts will be followed for survival every 2 mos after PD for up to 12 mos from the date of enrollment of the last pt.
To evaluate the safety profile of S-1 | Each cycle will last 21 days (14 days treatment, 7 days recovery) until death/removal from study. AEs reported through f/up; blood/urine collected at baseline, Days 8&15, w/in 24 hrs of drug on Day 1 of each cycle after Cycle 1, at end of treatment.
To investigate the relationship of S-1 plasma levels (components and metabolites) with safety and efficacy parameters | Each cycle will last 21 days (14 days treatment, 7 days recovery) until death or removal from study for any reason. s Blood samples to be obtained 1.5 ± 0.5 h, 5 ± 1 h, 7 ± 1 h postdose on Day 1 of Cycle 1 only.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Benedetti, MD, Study Director — Taiho Oncology, Inc.